CLINICAL TRIAL: NCT03840343
Title: Intra-arterially Delivered Autologous Mesenchymal Stem/Stromal Cell Therapy in Patients With Diabetic Kidney Disease: A Phase I Study
Brief Title: Patient-Derived Stem Cell Therapy for Diabetic Kidney Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator relocation
Sponsor: Mayo Clinic (Other)
Collaborators: Regenerative Medicine Minnesota (Unknown)
Responsible Party: Principal Investigator, LaTonya J. Hickson, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-002423; RMM 091718 CT 001 (Other Grant/Funding Number: Regenerative Medicine Minnesota)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Kidney Disease; Diabetic Nephropathies; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Chronic Kidney Disease; Diabetic Nephropathy Type 2; Kidney Failure; Kidney Insufficiency
Keywords: Mesenchymal Stem Cell; Mesencymal Stromal Cell; Stem Cell; Regenerative Medicine; Cell therapy; Rejuvenation
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower Dose MSC (Experimental): This arm will receive autologous adipose-derived Mesenchymal stem/stromal cells (MSC) Lower Dose.
  Interventions: Biological: Autologous adipose-derived mesenchymal stem/stromal cells (MSC) Lower Dose
- Higher Dose MSC (Experimental): This arm will receive autologous adipose-derived Mesenchymal stem/stromal cells (MSC) Higher Dose
  Interventions: Biological: Autologous adipose-derived mesenchymal stem/stromal cells (MSC) Higher Dose

INTERVENTIONS:
Biological: Autologous adipose-derived mesenchymal stem/stromal cells (MSC) Lower Dose — Two MSC infusions of 2.5x10^5 cells/kg at time zero and three months; single kidney, intra-arterial delivery
  Arms: Lower Dose MSC
Biological: Autologous adipose-derived mesenchymal stem/stromal cells (MSC) Higher Dose — Two MSC infusions of 5.0x10^5 cells/kg at time zero and three months; single kidney, intra-arterial delivery
  Arms: Higher Dose MSC

SUMMARY:
The Researchers will assess the safety, tolerability, dosing effect, and early signals of efficacy of intra-arterially delivered autologous (from self) adipose (fat) tissue-derived mesenchymal stem/stromal cells (MSC) in patients with progressive diabetic kidney disease (DKD).

DETAILED DESCRIPTION:
This is a single center, open-label dose-escalating study assessing safety, tolerability, dosing effect, and early signals of efficacy of intra-arterially delivered autologous (from self) adipose tissue-derived mesenchymal stem/stromal cells (MSC) in 30 patients with progressive diabetic kidney disease (DKD). DKD will be defined as chronic kidney disease (CKD; estimated glomerular filtration rate; eGFR<60 mL/min/1.73m2) in the setting of diabetes mellitus (type 2; on anti-diabetes therapy) without overt etiologies of CKD beyond concomitant hypertension. Progressive DKD will be considered as eGFR 25-55 ml/min/1.73m2 with a) eGFR decline of 5 ml/min over 18 months or 10 ml/min over 3 years or b) an intermediate or high 5-year risk of progression to end-stage kidney failure (dialysis or transplant) based on the validated Tangri 4-variable (age, sex, eGFR, urinary albumin-creatinine ratio) kidney failure risk equation. Fifteen subjects will be placed in one of two cell dosage arms in a parallel design with single-kidney MSC administration at Day 0 and Month 3. Subjects will be followed a total of 15 months from time of initial cell administration.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (on anti-diabetes drug therapy)
* Age 45-75 years
* eGFR 25-55 ml/min/1.73m2 at time of consent with: a) eGFR decline of 5 ml/min over 18 months or 10 ml/min over 3 years or b) an intermediate or high 5-year risk of progression to end-stage kidney failure (dialysis or transplant) based on the validated Tangri 4-variable (age, sex, eGFR, urinary albumin-creatinine ratio) kidney failure risk equation https://kidneyfailurerisk.com/
* Primary cause of kidney disease is diabetes without suspicion of concomitant kidney disease beyond hypertension
* Spot urine albumin:creatinine ≥30 mg/g unless on RAAS inhibition
* Ability to give informed consent

Exclusion Criteria:

* Hemoglobin A1c≥11%
* Pregnancy
* Active malignancy
* Active Immunosuppression therapy
* Kidney transplantation history
* Concomitant glomerulonephritis
* Nephrotic syndrome
* Solid organ transplantation history
* Autosomal dominant or recessive polycystic kidney disease
* Known renovascular disease
* Kidney failure (hemodialysis, peritoneal dialysis, or kidney transplantation)
* Active tobacco use
* Body weight >150 kg or BMI>50
* Uncontrolled hypertension: Systolic blood pressure (SBP) >180 mmHg despite antihypertensive therapy
* Recent cardiovascular event (myocardial infarction, stroke, congestive heart failure within 6 months
* Evidence of hepatitis B or C, or HIV infection, chronic
* Anticoagulation therapy requiring heparin bridging for procedures.
* History of methicillin-resistant staphylococcus aureus colonization
* Recent plastic, chemical or surgical manipulation of adipose tissue for cosmetic purposes within 6 months
* Inability to give informed consent
* Potentially unreliable subjects and those judged by the investigator to be unsuitable for the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Baseline through Month 15
  The number of Adverse Events associated with MSC intervention per treatment arm
Adverse Events | Baseline through Month 15
  The percentage of Adverse Events associated with MSC intervention per treatment arm

SECONDARY OUTCOMES:
Kidney Function | baseline, month 6
  Change in measured glomerular filtration rate (mGFR). Measured as mL/min/BSA
Kidney Function | pretreatment, month 12
  Change in estimated glomerular filtration rate (eGFR) slope. Measured as mL/min/1.73m^2/month

CONTACTS AND LOCATIONS:
Overall Officials: LaTonya J Hickson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alatta LS, Elhusseiny KM, Dietz AB, Herrmann SM, Lorenz EC, Lawson DK, Bendel EC, Reisenauer CJ, Misra S, Vaughan LE, Lerman LO, Hickson LJ. Intraarterial Autologous Mesenchymal Stem Cell Therapy for Diabetic Kidney Disease. Kidney Int Rep. 2025 Aug 6;10(10):3656-3660. doi: 10.1016/j.ekir.2025.07.042. eCollection 2025 Oct. No abstract available. PMID 41141513
- [Background] Patel HA, Wang J, Zinn CJ, Learmonth M, Lerman LO, Wolfram J, Hickson LJ. Fortifying the Diabetic Kidney Disease Treatment Armamentarium: Multitarget Senotherapeutic and Regenerative Strategies. J Am Soc Nephrol. 2025 May 7;36(8):1655-1658. doi: 10.1681/ASN.0000000754. No abstract available. PMID 40333016
- See also: Diabetic Kidney Disease Stem Cell Trial - Mayo Clinic — https://www.mayo.edu/research/clinical-trials/cls-20438442
- See also: Video of Stem Cell Trial in Diabetic Kidney Disease - Regenerative Medicine Minnesota — https://youtu.be/DQ7r3UFMDN8